CLINICAL TRIAL: NCT06088329
Title: Mindfulness Walking for Adults With Chronic Pain
Brief Title: Mindful Walking for Adults With Chronic Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clemson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB2023-0240
Record Dates: First submitted 2023-10-04; First posted 2023-10-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindful Walking (Experimental): All participants will belong to the experimental mindful walking arm for our single arm feasibility study.
  Interventions: Behavioral: Mindful Walking for Adults with Chronic Pain

INTERVENTIONS:
Behavioral: Mindful Walking for Adults with Chronic Pain — Participants identified with chronic pain will complete 6 sessions of mindfulness based walking exercises.

SUMMARY:
Both mindfulness-based interventions and light physical activity have been shown as effective in reducing the burden of chronic pain. This proposed intervention, mindful walking (MW), is a combination of physical activity and mindfulness-based intervention aimed at reducing pain with a non-pharmacological approach. In MW, mindfulness-based instructions emphasized acknowledging arising thoughts, feelings, and/or emotions without judgment or emotional reaction and to "simply return their attention back to the footstep" sensation whenever such discursive events occur. Furthermore, subjects will be taught that perceived sensory and affective events were "momentary" and "fleeting" and do not require further interpretation or evaluation.

DETAILED DESCRIPTION:
Specifically, our proposed MW intervention will focus on the following:

1. Participants will be instructed to focus on the sensations occurring "at the toes or at sole."
2. Participants will be instructed to expand their focus to the "full length of the step," including bodily sensations (e.g., rise and fall of the abdomen and chest).
3. Participants will learn the application of mindfulness principles with the goal for use in everyday life.

The anticipation is to include thirty patients in Clemson South Carolina with chronic pain without any prior meditative experience (diabetes patients with neuropathic pain, prostate cancer patients with postoperative pain, etc.) into our study.

Eligible participants will then complete 6 sessions of mindful walking across 6 weeks. Each weekly session will last approximately 60 minutes and will be conducted outdoors (weather pending). Mindful walking is a practice of becoming aware of one's surroundings and internal feelings while moving. When practicing walking mindfully, one focuses his/her attention on the sensations in the body with each step, paying close attention to the breath. The mindful walking sessions are intended to provide therapeutic techniques based on achieving a state of mind that focuses one's awareness on the present moment while acknowledging and accepting one's thoughts/feelings. Sessions will be led by a certified instructor to follow mindfulness practices with the incorporation of walking for adults with chronic pain.

At the end of the sessions, participants will be randomly selected using a random number generator to participate in an informal interview session. This is an opportunity for participants to tell us about their experiences in the program and how mindful walking has impacted their chronic pain. The interview will take about thirty minutes of their time.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years of age or older
* Residents in Oconee and Pickens County
* Individuals with mild to severe chronic pain (i.e., neuropathic pain, postoperative pain, migraine headaches, etc.)
* Individuals must be able to read and understand English (can speak other languages), a translator will not be provided.

Exclusion Criteria:

* Current Mindfulness practice.
* Individuals without chronic pain.
* Individuals who cannot walk without assistance for more than 5 minutes.
* Individuals who do not experience mild to severe chronic pain for at least 3 days per week every week on average.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-11-14 (Actual); Primary Completion 2023-12-06 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Over a 6 week time frame from the start at baseline of the study (week 0) to the end of the study (week 6).
  Measure participants perceived level of pain using validated scales Brief Pain Inventory for pain level 0 meaning no pain and 10 meaning pain as bad as you can imagine.
Unpleasantness of the pain | Over a 6 week time frame from the start at baseline of the study (week 0) to the end of the study (week 6).
  Understand participants perceived level of pain using questionnaire Brief Pain Inventory for pain level 0 meaning no pain and 10 meaning pain as bad as you can imagine and qualitative responses.
Pain-related functional scale | Over a 6 week time frame from the start at baseline of the study (week 0) to the end of the study (week 6).
  Measure participants perceived level of pain using validated scales for pain level (Visual Pain scale 0 meaning no pain and 10 being the worst pain.
Pain-related quality of life | Over a 6 week time frame from the start at baseline of the study (week 0) to the end of the study (week 6).
  Understand participants perceived level of pain using validated scales for pain level (Visual Pain scale Pain scale 0 meaning no pain and 10 being the worst pain. Also use qualitative data responses.

SECONDARY OUTCOMES:
Mindfulness inventory | Over a 6 week time frame from the start at baseline of the study (week 0) to the end of the study (week 6).
  Assess the effect of mindfulness techniques based on survey questions and qualitative responses.
Perceived intervention effectiveness of pain change | Over a 6 week time frame from the start at baseline of the study (week 0) to the end of the study (week 6).
  Perceived intervention effectiveness of pain change will be assessed with a Visual Analogue Scale (VAS) ("0" = not effective at all; "10"= most effective imaginable, for each intervention session's assigned intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lu Shi, Principal Investigator — Clemson University
Locations (1):
- Clemson University, Clemson, South Carolina, United States